CLINICAL TRIAL: NCT06416462
Title: Action of Photodynamic Therapy on Wound Quality and Tissue Repair in the Diabetic Foot: Double Blind Randomized Controlled Clinical Study
Brief Title: Action of Photodynamic Therapy on Wound Quality and Tissue Repair in the Diabetic Foot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Kristianne Porta Santos Fernandes, Clinical colaborator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6.296.354
Record Dates: First submitted 2023-10-02; First posted 2024-05-16 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simulation of antimicroial Photodynamic therapy group (Placebo Comparator): Participants in the control group will be treated in exactly the same way as the aPDT group, however the light treatment will be simulated. The device will be placed in position, however it will be switched off. After three weeks of monitoring in the control group, the patient will be informed that they were in the placebo group and will be offered treatment with aPDT and irradiation, for ethical reasons.
  Interventions: Procedure: antimicrobial photodynamic therapy
- Antimicrobial Photodynamic therapy group (Active Comparator): In the experimental group (aPDT), 1% methylene blue applied with the aid of a syringe will be used as a photosensitizer (with a pre-irradiation time of 5 minutes, 6 J of red laser will be applied.
  Interventions: Procedure: antimicrobial photodynamic therapy

INTERVENTIONS:
Procedure: antimicrobial photodynamic therapy — When starting the research, all wounds, regardless of the study group, will be cleaned with 0.9% saline solution (SF0.9%), using a 40x12 needle and a 500ml bottle of SF0.9%, in order to maintain pressure. for equal cleaning of all wounds and a hydrofiber plate with silver was used as standard coverage. Experimental group (n=45): When starting the intervention, all services in both groups will follow the cleaning standard described previously. In the aPDT group, 1% methylene blue will be used as a photosensitizer applied with the aid of a syringe (with a pre-irradiation time of 5 minutes), 6 J of laser will be applied.

SUMMARY:
Diabetic foot ulcer affects 10.5% of the Brazilian/world population, compromising the quality of life of these patients and burdening the public health system. Studies show that antimicrobial photodynamic therapy (aPDT) accelerates its repair, however, there is not enough evidence for decision-making in clinical practice, which prevents this treatment from being used on a large scale. Controlled and randomized clinical studies are needed to increase the level of evidence on this subject, promoting the improvement of the quality of life of people affected by diabetic foot ulcers. The aim of this study is to analyze the action of antimicrobial photodynamic therapy on the quality of the wound and tissue repair process using the Bates-Jensen scale in people affected by diabetic foot wounds.

DETAILED DESCRIPTION:
Diabetic foot ulcer affects 10.5% of the Brazilian/world population, compromising the quality of life of these patients and burdening the public health system. Studies show that antimicrobial photodynamic therapy (aPDT) accelerates its repair, however, there is not enough evidence for decision-making in clinical practice, which prevents this treatment from being used on a large scale. Controlled and randomized clinical studies are needed to increase the level of evidence on this subject, promoting the improvement of the quality of life of people affected by diabetic foot ulcers. The aim of this study is to analyze the action of antimicrobial photodynamic therapy on the quality of the wound and tissue repair process using the Bates-Jensen scale in people affected by diabetic foot wounds. A clinical, controlled, randomized and double-blind study will be carried out. Patients will be randomized (1:1) into 2 groups: (1) experimental (n= 45) - standard care from the Polyclinic wound sector + aPDT and (2) control (n= 45) - standard care + simulation of use aPDT with equipment off). All patients will be seen three times a week, with 10 sessions of aPDT or simulation performed by the same operator. A cluster with an average radiant power of 100 mW, radiant energy per emitter of 6 J/cm² of red light (wavelength 660 nm) will be used. The research will be carried out in a Municipal Health Center in the city of Rio de Janeiro. Patients affected by neuropathic wounds of the diabetic foot, assisted by the Programmatic Care Health Coordination will be included 5.1. The initial assessment will consist of collecting data from medical records to establish the sociodemographic and clinical profile of patients affected by diabetic foot injuries.) by a researcher blinded to the interventions. This scale assesses the size of the lesion, depth, borders, detachment, type of necrotic tissue, amount of necrotic tissue, type of exudate, amount of exudate, skin color around the wound, perilesional tissue edema, perilesional tissue hardening, granulation tissue, epithelialization. As secondary outcomes: the sensitivity of the foot will be evaluated, through neurological evaluation with tuning fork and monofilament, the instrument for assessing quality of life - Diabetes-21, the Wagner Scale, the evaluation of the degree of ischemia by the Fontaine scale and Runtherford, the WiFi and Taxonomy Nursing Outcomes Classification scale that assesses skin integrity. Data from this research will be collected after approval by the ethics committee of Universidade Nove de Julho and the City Hall of Rio de Janeiro.

ELIGIBILITY:
Inclusion Criteria:

* both sexes
* chronic wounds originating from the neuropathic diabetic foot
* contaminated lesions
* total score obtained on the Bates-Jensen scale between 13 and 60
* who submits all requested exams

Exclusion Criteria:

* wounds with etiologies that are not related to the diabetic foot
* ischemic diabetic foot who has an ankle-brachial index with a value between 0.7 and 1.3.
* glycated hemoglobin greater than 8%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Bates-Jensen Wound Assesment Tool | Before the intervention
  The Bates-Jensen Scale is an effective tool for wound assessment. In its current version, it includes 13 characteristics to be evaluated: size, depth, edges, undermining, type of necrotic tissue, amount of necrotic tissue, exudate type, exudate amount, skin color around the wound, perilesional tissue edema, perilesional tissue induration, granulation tissue, and epithelialization.
  Each item on the scale is scored from 1 to 5:
  minimum values indicate the best wound condition,
  maximum values represent the worst condition.
  The total score is obtained by summing all the items and can range from 13 to 65 points, with HIGHER scores indicating WORSE wound conditions.
Bates-Jensen Wound Assesment Tool | First day after intervention
  The Bates-Jensen Scale is an effective tool for wound assessment. In its current version, it includes 13 characteristics to be evaluated: size, depth, edges, undermining, type of necrotic tissue, amount of necrotic tissue, exudate type, exudate amount, skin color around the wound, perilesional tissue edema, perilesional tissue induration, granulation tissue, and epithelialization.
  Each item on the scale is scored from 1 to 5:
  minimum values indicate the best wound condition,
  maximum values represent the worst condition.
  The total score is obtained by summing all the items and can range from 13 to 65 points, with HIGHER scores indicating WORSE wound conditions.
Bates-Jensen scale | Third day after intervention
  The Bates-Jensen Scale is an effective tool for wound assessment. In its current version, it includes 13 characteristics to be evaluated: size, depth, edges, undermining, type of necrotic tissue, amount of necrotic tissue, exudate type, exudate amount, skin color around the wound, perilesional tissue edema, perilesional tissue induration, granulation tissue, and epithelialization.
  Each item on the scale is scored from 1 to 5:
  minimum values indicate the best wound condition,
  maximum values represent the worst condition.
  The total score is obtained by summing all the items and can range from 13 to 65 points, with HIGHER scores indicating WORSE wound conditions.
Bates-Jensen scale | Fifth day after intervention
  The Bates-Jensen Scale is an effective tool for wound assessment. In its current version, it includes 13 characteristics to be evaluated: size, depth, edges, undermining, type of necrotic tissue, amount of necrotic tissue, exudate type, exudate amount, skin color around the wound, perilesional tissue edema, perilesional tissue induration, granulation tissue, and epithelialization.
  Each item on the scale is scored from 1 to 5:
  minimum values indicate the best wound condition,
  maximum values represent the worst condition.
  The total score is obtained by summing all the items and can range from 13 to 65 points, with HIGHER scores indicating WORSE wound conditions.
Bates-Jensen scale | Tenth day after intervention
  The Bates-Jensen Scale is an effective tool for wound assessment. In its current version, it includes 13 characteristics to be evaluated: size, depth, edges, undermining, type of necrotic tissue, amount of necrotic tissue, exudate type, exudate amount, skin color around the wound, perilesional tissue edema, perilesional tissue induration, granulation tissue, and epithelialization. Each item on the scale is scored from 1 to 5, where 1 indicates the best wound condition, and 5 represents the worst condition. The total score is obtained by summing all the items and can range from 13 to 65 points, with higher scores indicating worse wound conditions.

SECONDARY OUTCOMES:
Diabetes twenty-one instrument | Before the intervention
  The Diabetes-21 (D-21) instrument evaluates the quality of life of individuals living with diabetes by assessing the condition's physical, emotional, and social impacts. It consists of 21 items scored on a Likert scale, reflecting the intensity or frequency of diabetes-related challenges. The scoring ranges from a minimum of 21 to a maximum of 105. Lower scores indicate a better quality of life, suggesting fewer diabetes-related difficulties, while higher scores reflect a worse quality of life, indicating more significant challenges or negative impacts. This makes the D-21 a valuable tool for assessing the burden of diabetes in both clinical and research settings.
Diabetes twenty-one instrument | First day after intervention
  he Diabetes-21 (D-21) instrument evaluates the quality of life of individuals living with diabetes by assessing the physical, emotional, and social impacts of the condition. It consists of 21 items scored on a Likert scale, reflecting the intensity or frequency of diabetes-related challenges. The scoring ranges from a minimum of 21 to a maximum of 105. Lower scores indicate a better quality of life, suggesting fewer diabetes-related difficulties, while higher scores reflect a worse quality of life, indicating more significant challenges or negative impacts. This makes the D-21 a valuable tool for assessing the burden of diabetes in both clinical and research settings.
Diabetes twenty-one instrument | Third day after intervention
  he Diabetes-21 (D-21) instrument evaluates the quality of life of individuals living with diabetes by assessing the physical, emotional, and social impacts of the condition. It consists of 21 items scored on a Likert scale, reflecting the intensity or frequency of diabetes-related challenges. The scoring ranges from a minimum of 21 to a maximum of 105. Lower scores indicate a better quality of life, suggesting fewer diabetes-related difficulties, while higher scores reflect a worse quality of life, indicating more significant challenges or negative impacts. This makes the D-21 a valuable tool for assessing the burden of diabetes in both clinical and research settings.
Diabetes twenty-one instrument | The fifth day after intervention
  he Diabetes-21 (D-21) instrument evaluates the quality of life of individuals living with diabetes by assessing the physical, emotional, and social impacts of the condition. It consists of 21 items scored on a Likert scale, reflecting the intensity or frequency of diabetes-related challenges. The scoring ranges from a minimum of 21 to a maximum of 105. Lower scores indicate a better quality of life, suggesting fewer diabetes-related difficulties, while higher scores reflect a worse quality of life, indicating more significant challenges or negative impacts. This makes the D-21 a valuable tool for assessing the burden of diabetes in both clinical and research settings.
Diabetes twenty-one instrument | Tenth day after intervention
  he Diabetes-21 (D-21) instrument evaluates the quality of life of individuals living with diabetes by assessing the physical, emotional, and social impacts of the condition. It consists of 21 items scored on a Likert scale, reflecting the intensity or frequency of diabetes-related challenges. The scoring ranges from a minimum of 21 to a maximum of 105. Lower scores indicate a better quality of life, suggesting fewer diabetes-related difficulties, while higher scores reflect a worse quality of life, indicating more significant challenges or negative impacts. This makes the D-21 a valuable tool for assessing the burden of diabetes in both clinical and research settings.
Wagner Scale | Before the intervention
  The Wagner Scale is a classification system used to evaluate the severity of diabetic foot ulcers. It categorizes ulcers based on depth, tissue involvement, and the presence of infection or gangrene. The scale ranges from 0 to 5, with higher scores indicating more severe conditions. A score of 0 represents a pre-ulcerative lesion or intact skin, while a score of 5 indicates extensive gangrene involving the entire foot. The Wagner Scale is widely used in clinical settings to guide treatment decisions and monitor the progression of diabetic foot complications.
Wagner Scale | First day after intervention
  The Wagner Scale is a classification system used to evaluate the severity of diabetic foot ulcers. It categorizes ulcers based on depth, tissue involvement, and the presence of infection or gangrene. The scale ranges from 0 to 5, with higher scores indicating more severe conditions. A score of 0 represents a pre-ulcerative lesion or intact skin, while a score of 5 indicates extensive gangrene involving the entire foot. The Wagner Scale is widely used in clinical settings to guide treatment decisions and monitor the progression of diabetic foot complications.
Wagner Scale | Third day after intervention
  The Wagner Scale is a classification system used to evaluate the severity of diabetic foot ulcers. It categorizes ulcers based on depth, tissue involvement, and the presence of infection or gangrene. The scale ranges from 0 to 5, with higher scores indicating more severe conditions. A score of 0 represents a pre-ulcerative lesion or intact skin, while a score of 5 indicates extensive gangrene involving the entire foot. The Wagner Scale is widely used in clinical settings to guide treatment decisions and monitor the progression of diabetic foot complications.
Wagner Scale | Fifth day after intervention
  The Wagner Scale is a classification system used to evaluate the severity of diabetic foot ulcers. It categorizes ulcers based on depth, tissue involvement, and the presence of infection or gangrene. The scale ranges from 0 to 5, with higher scores indicating more severe conditions. A score of 0 represents a pre-ulcerative lesion or intact skin, while a score of 5 indicates extensive gangrene involving the entire foot. The Wagner Scale is widely used in clinical settings to guide treatment decisions and monitor the progression of diabetic foot complications.
Wagner Scale | Tenth day after intervention
  The Wagner Scale is a classification system used to evaluate the severity of diabetic foot ulcers. It categorizes ulcers based on depth, tissue involvement, and the presence of infection or gangrene. The scale ranges from 0 to 5, with higher scores indicating more severe conditions. A score of 0 represents a pre-ulcerative lesion or intact skin, while a score of 5 indicates extensive gangrene involving the entire foot. The Wagner Scale is widely used in clinical settings to guide treatment decisions and monitor the progression of diabetic foot complications.
WiFi scale | Before the intervention
  The WiFi scale is a classification system used to assess the severity of diabetic foot ulcers by evaluating three key factors: wound size and depth (W), ischemia (I), and foot infection (Fi). Each component is graded from 0 to 3, with higher grades indicating more severe conditions. The combined scores help determine the overall risk of amputation and guide treatment planning. A higher overall score indicates a worse prognosis and increased need for advanced interventions. The WiFi scale is widely used in clinical practice to stratify risk and optimize care for patients with diabetic foot complications.
WiFi scale | First day after intervention
  The WiFi scale is a classification system used to assess the severity of diabetic foot ulcers by evaluating three key factors: wound size and depth (W), ischemia (I), and foot infection (Fi). Each component is graded from 0 to 3, with higher grades indicating more severe conditions. The combined scores help determine the overall risk of amputation and guide treatment planning. A higher overall score indicates a worse prognosis and increased need for advanced interventions. The WiFi scale is widely used in clinical practice to stratify risk and optimize care for patients with diabetic foot complications.
WiFi scale | Third day after intervention
  The WiFi scale is a classification system used to assess the severity of diabetic foot ulcers by evaluating three key factors: wound size and depth (W), ischemia (I), and foot infection (Fi). Each component is graded from 0 to 3, with higher grades indicating more severe conditions. The combined scores help determine the overall risk of amputation and guide treatment planning. A higher overall score indicates a worse prognosis and increased need for advanced interventions. The WiFi scale is widely used in clinical practice to stratify risk and optimize care for patients with diabetic foot complications.
WiFi scale | Fifth day after intervention
  The WiFi scale is a classification system used to assess the severity of diabetic foot ulcers by evaluating three key factors: wound size and depth (W), ischemia (I), and foot infection (Fi). Each component is graded from 0 to 3, with higher grades indicating more severe conditions. The combined scores help determine the overall risk of amputation and guide treatment planning. A higher overall score indicates a worse prognosis and increased need for advanced interventions. The WiFi scale is widely used in clinical practice to stratify risk and optimize care for patients with diabetic foot complications.
WiFi scale | Tenth day after intervention
  The WiFi scale is a classification system used to assess the severity of diabetic foot ulcers by evaluating three key factors: wound size and depth (W), ischemia (I), and foot infection (Fi). Each component is graded from 0 to 3, with higher grades indicating more severe conditions. The combined scores help determine the overall risk of amputation and guide treatment planning. A higher overall score indicates a worse prognosis and increased need for advanced interventions. The WiFi scale is widely used in clinical practice to stratify risk and optimize care for patients with diabetic foot complications.
Nursing Outcomes Classification Taxonomy | Before the intervention
  Assess skin integrity using the Nursing Outcomes Classification Taxonomy
Nursing Outcomes Classification Taxonomy | First day after intervention
  Assess skin integrity using the Nursing Outcomes Classification Taxonomy
Nursing Outcomes Classification Taxonomy | Third day after intervention
  Assess skin integrity using the Nursing Outcomes Classification Taxonomy
Nursing Outcomes Classification Taxonomy | Fifth day after intervention
  Assess skin integrity using the Nursing Outcomes Classification Taxonomy
Nursing Outcomes Classification Taxonomy | Tenth day after intervention
  Assess skin integrity using the Nursing Outcomes Classification Taxonomy
Runtherford Scale for ischemia evaluation | Before the intervention
  Classification on the degree of ischemia, with some differences in the parameters assessed: asymptomatic (0); mild claudication (1); moderate claudication (2); severe claudication (3); ischemic pain at rest (4); minor tissue loss (5); major tissue loss (6). The higher value corresponds to the worst result.
Runtherford Scale for ischemia evaluation | First day after intervention
  Classification on the degree of ischemia, with some differences in the parameters assessed: asymptomatic (0); mild claudication (1); moderate claudication (2); severe claudication (3); ischemic pain at rest (4); minor tissue loss (5); major tissue loss (6). The higher value corresponds to the worst result.
Runtherford Scale for ischemia evaluation | Third day after intervention
  Classification on the degree of ischemia, with some differences in the parameters assessed: asymptomatic (0); mild claudication (1); moderate claudication (2); severe claudication (3); ischemic pain at rest (4); minor tissue loss (5); major tissue loss (6). The higher value corresponds to the worst result.
Runtherford Scale for ischemia evaluation | Fifth day after intervention
  Classification on the degree of ischemia, with some differences in the parameters assessed: asymptomatic (0); mild claudication (1); moderate claudication (2); severe claudication (3); ischemic pain at rest (4); minor tissue loss (5); major tissue loss (6). The higher value corresponds to the worst result.
Runtherford Scale for ischemia evaluation | Tenth day after intervention
  Classification on the degree of ischemia, with some differences in the parameters assessed: asymptomatic (0); mild claudication (1); moderate claudication (2); severe claudication (3); ischemic pain at rest (4); minor tissue loss (5); major tissue loss (6). The higher value corresponds to the worst result.
protective sensitivity of the feet through the monofilament | Before the intervention
  The protective sensitivity test using a monofilament evaluates whether an individual can feel pressure on specific points of their feet. The outcome is classified as either the presence or absence of protective sensation.
protective sensitivity of the feet through the monofilament | First day after intervention
  The protective sensitivity test using a monofilament evaluates whether an individual can feel pressure on specific points of their feet. The outcome is classified as either the presence or absence of protective sensation.
protective sensitivity of the feet through the monofilament | Third day after intervention
  The protective sensitivity test using a monofilament evaluates whether an individual can feel pressure on specific points of their feet. The outcome is classified as either the presence or absence of protective sensation.
protective sensitivity of the feet through the monofilament | Fifth day after intervention
  The protective sensitivity test using a monofilament evaluates whether an individual can feel pressure on specific points of their feet. The outcome is classified as either the presence or absence of protective sensation.
protective sensitivity of the feet through the monofilament | Tenth day after intervention
  The protective sensitivity test using a monofilament evaluates whether an individual can feel pressure on specific points of their feet. The outcome is classified as either the presence or absence of protective sensation.
protective sensitivity of the feet through tuning fork test | Before the intervention
  The protective sensitivity test using a tuning fork evaluates the ability to perceive vibration in specific points on the feet, typically at bony prominences. The outcome is classified as either the presence or absence of protective sensation.
protective sensitivity of the feet through tuning fork test | First day after intervention
  The protective sensitivity test using a tuning fork evaluates the ability to perceive vibration in specific points on the feet, typically at bony prominences. The outcome is classified as either the presence or absence of protective sensation.
protective sensitivity of the feet through tuning fork test | Third day after intervention
  The protective sensitivity test using a tuning fork evaluates the ability to perceive vibration in specific points on the feet, typically at bony prominences. The outcome is classified as either the presence or absence of protective sensation.
protective sensitivity of the feet through tuning fork test | Fifth day after intervention
  The protective sensitivity test using a tuning fork evaluates the ability to perceive vibration in specific points on the feet, typically at bony prominences. The outcome is classified as either the presence or absence of protective sensation.
protective sensitivity of the feet through tuning fork test | Tenth day after intervention
  The protective sensitivity test using a tuning fork evaluates the ability to perceive vibration in specific points on the feet, typically at bony prominences. The outcome is classified as either the presence or absence of protective sensation.
Fontaine Classification | Before the intervention
  primarily rely on the degree of limb ischemia, evaluating the following parameters: asymptomatic (I); mild claudication (IIa); moderate to severe claudication (IIb); rest pain (III); gangrene or ulceration (IV).
Fontaine Classification | First day after intervention
  primarily rely on the degree of limb ischemia, evaluating the following parameters: asymptomatic (I); mild claudication (IIa); moderate to severe claudication (IIb); rest pain (III); gangrene or ulceration (IV).
Fontaine Classification | Third day after intervention
  primarily rely on the degree of limb ischemia, evaluating the following parameters: asymptomatic (I); mild claudication (IIa); moderate to severe claudication (IIb); rest pain (III); gangrene or ulceration (IV).
Fontaine Classification | Fifth day after intervention
  primarily rely on the degree of limb ischemia, evaluating the following parameters: asymptomatic (I); mild claudication (IIa); moderate to severe claudication (IIb); rest pain (III); gangrene or ulceration (IV).
Fontaine Classification | Tenth day after intervention
  primarily rely on the degree of limb ischemia, evaluating the following parameters: asymptomatic (I); mild claudication (IIa); moderate to severe claudication (IIb); rest pain (III); gangrene or ulceration (IV).
Vibration Sensation | Before the intervention
  To assess vibratory sensitivity, a 128Hz tuning fork is applied to a bony area (e.g., elbow, clavicle, sternum, chin) to demonstrate the expected sensation. The participant then closes their eyes, and the tuning fork is applied with constant pressure to the dorsal side of the hallux's distal phalanx or another toe if the hallux is missing. If all phalanges are amputated, it's applied to the nearby area. The tuning fork is held in place until the participant reports the vibration has ceased. The test is repeated twice, with at least one "simulated" application where the tuning fork doesn't vibrate. A positive test result is when the participant correctly identifies vibration in at least two out of three applications, while a negative result is when they inaccurately identify vibration in two out of three applications, indicating a lack of vibratory sensitivity
Vibration Sensation | First day after intervention
  To assess vibratory sensitivity, a 128Hz tuning fork is applied to a bony area (e.g., elbow, clavicle, sternum, chin) to demonstrate the expected sensation. The participant then closes their eyes, and the tuning fork is applied with constant pressure to the dorsal side of the hallux's distal phalanx or another toe if the hallux is missing. If all phalanges are amputated, it's applied to the nearby area. The tuning fork is held in place until the participant reports the vibration has ceased. The test is repeated twice, with at least one "simulated" application where the tuning fork doesn't vibrate. A positive test result is when the participant correctly identifies vibration in at least two out of three applications, while a negative result is when they inaccurately identify vibration in two out of three applications, indicating a lack of vibratory sensitivity
Vibration Sensation | Third day after intervention
  To assess vibratory sensitivity, a 128Hz tuning fork is applied to a bony area (e.g., elbow, clavicle, sternum, chin) to demonstrate the expected sensation. The participant then closes their eyes, and the tuning fork is applied with constant pressure to the dorsal side of the hallux's distal phalanx or another toe if the hallux is missing. If all phalanges are amputated, it's applied to the nearby area. The tuning fork is held in place until the participant reports the vibration has ceased. The test is repeated twice, with at least one "simulated" application where the tuning fork doesn't vibrate. A positive test result is when the participant correctly identifies vibration in at least two out of three applications, while a negative result is when they inaccurately identify vibration in two out of three applications, indicating a lack of vibratory sensitivity
Vibration Sensation | Fifth day after intervention
  To assess vibratory sensitivity, a 128Hz tuning fork is applied to a bony area (e.g., elbow, clavicle, sternum, chin) to demonstrate the expected sensation. The participant then closes their eyes, and the tuning fork is applied with constant pressure to the dorsal side of the hallux's distal phalanx or another toe if the hallux is missing. If all phalanges are amputated, it's applied to the nearby area. The tuning fork is held in place until the participant reports the vibration has ceased. The test is repeated twice, with at least one "simulated" application where the tuning fork doesn't vibrate. A positive test result is when the participant correctly identifies vibration in at least two out of three applications, while a negative result is when they inaccurately identify vibration in two out of three applications, indicating a lack of vibratory sensitivity
Vibration Sensation | Tenth day after intervention
  To assess vibratory sensitivity, a 128Hz tuning fork is applied to a bony area (e.g., elbow, clavicle, sternum, chin) to demonstrate the expected sensation. The participant then closes their eyes, and the tuning fork is applied with constant pressure to the dorsal side of the hallux's distal phalanx or another toe if the hallux is missing. If all phalanges are amputated, it's applied to the nearby area. The tuning fork is held in place until the participant reports the vibration has ceased. The test is repeated twice, with at least one "simulated" application where the tuning fork doesn't vibrate. A positive test result is when the participant correctly identifies vibration in at least two out of three applications, while a negative result is when they inaccurately identify vibration in two out of three applications, indicating a lack of vibratory sensitivity

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Agnelli Mesquita-Ferrari, PhD, Study Director — University of Nove de Julho
Locations (1):
- Raquel Agnelli Mesquita-Ferrari, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Chagas PF, Dos Santos TB, Dos Santos Trivino G, Bussadori SK, Duran CCG, Fernandes KPS, Cecatto RB, Horliana ACRT, Mesquita-Ferrari RA. Antimicrobial Photodynamic Therapy in Diabetic Amputation Ulcers: Case Series Evaluating Wound Healing Quality. Lasers Surg Med. 2025 Aug;57(6):457-465. doi: 10.1002/lsm.70037. Epub 2025 Jun 22. PMID 40545698